CLINICAL TRIAL: NCT01160328
Title: Influence of Male Hormones on Regional Fat Metabolism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Abbott (Industry)
Responsible Party: Principal Investigator, Michael D. Jensen, Michael D. Jensen, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 09-000309; R01DK045343 (NIH)
Record Dates: First submitted 2010-07-08; First posted 2010-07-12 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Obesity
Keywords: Regional Fat Storage; Fat Oxidation; Testosterone; Male
MeSH Terms: conditions — Obesity | interventions — Leuprolide; Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Group (No Intervention): Participants in this group will not receive any treatment.
- Lupron Group (Experimental): Participants in this group will receive leuprolide acetate (Lupron) treatment for 7 weeks resulting in temporary decreases in testosterone levels.
  Interventions: Drug: Leuprolide
- Lupron & Testosterone Group (Other): Participants in this group will receive 7 weeks of leuprolide acetate (Lupron) treatment with testosterone gel (Androgel).
  Interventions: Drug: Leuprolide; Drug: Testosterone

INTERVENTIONS:
Drug: Leuprolide — 7.5 mg - 1 month depot, 2 doses over 7 weeks
  Other Names: Lupron
  Arms: Lupron & Testosterone Group; Lupron Group
Drug: Testosterone — 7.5g - 1% testosterone gel, daily x 7 weeks
  Other Names: AndroGel
  Arms: Lupron & Testosterone Group

SUMMARY:
The male sex hormone, testosterone, plays an important role in determining body fat distribution in men. This is especially evident in the dramatic shift in body composition as boys and girls reach sexual maturity. Normal weight women have twice the body fat of a normal weight man (30% vs. 15% on average) and men will have twice the stomach fat as women (10% vs. 5% of fat as intra-abdominal, men vs. women). These are likely sex-steroid linked events. Short and long term changes in regional fat distribution accompany testosterone deficiency and can be reversed by testosterone replacement. Testosterone deficient men have increased stomach fat that can be reversed with testosterone replacement therapy. Interestingly, the mechanism by which testosterone affects where we store fat is unknown. It is important to understand how testosterone influences where we store fat as it is well established that increased stomach fat results in elevated disease risk.

The proposed study aims to examine the effect of short term, temporary testosterone decreases on how and where men store fat. The investigators will compare fat storage between men given Lupron to temporarily decrease testosterone levels those that receive Lupron plus testosterone replacement vs. a no treatment control group. Comparing these three groups will allow us to understand the effects of testosterone on short-term changes in fat tissue function that lead to the long-term changes in where we store body fat.

DETAILED DESCRIPTION:
There are 3 groups to which you might be assigned. Assignment to these groups is random (ie. by flip of a coin).

If you are assigned to…

* Group 1 - you will receive no treatments.
* Group 2 - you will be given an injection of leuprolide acetate (Lupron) which will temporarily lower sex hormones. This injection will be given two times during the 7 week treatment period.
* Group 3 - you will be given the injections of Lupron but after the second injection, you will also be required to apply a testosterone gel that will result in maintenance of your testosterone levels. The testosterone gel is rubbed on the upper shoulders, similar to putting on suntan lotion. You will be shown how to put this on.

If you are in group 2 or 3 you will be given testosterone gel, a male hormone, at the end of the study to help prevent symptoms such as hot flashes, until your body has time to return to its pre-study hormone levels. This can take up to 4 weeks.

In addition to the treatment period, you will also:

* If you are in group 1, have 4 fat biopsies that are like a miniature liposuction. The investigators numb the skin before doing the biopsies. If you are in group 2 or 3, you will also have 1 muscle biopsy at the end of the treatment period. In addition, if you are in group 2 or 3, you will also have a fat and muscle biopsy before you start the hormone treatment.
* All groups will need to spend two days and nights in the Clinical Research Unit of the Mayo Clinic and your meals will be provided by the for 5 days beforehand. You will also need to spend one morning undergoing some initial tests.
* You will have your body fat measured before and after the hormone treatment using x-ray like equipment that will expose you to some radiation.
* Our measures of fat metabolism use molecules that have a small amount of radioactivity.

Remuneration is provided.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, weight stable individuals
* BMI 20-29 kg/m2

Exclusion Criteria:

* Smoking and tobacco use
* Diabetes and other disease
* Anti-depressants

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2010-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Regional Fat Metabolism | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Jensen, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States